CLINICAL TRIAL: NCT02693860
Title: A Pilot Study of Neoadjuvant Monoclonal Antibody Humanised (hu) J591 for the Treatment of High and/or Intermediate-Risk Prostate Cancer
Brief Title: Neoadjuvant J591 Treatment for Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1505016234
Record Dates: First submitted 2016-02-12; First posted 2016-02-29 (Estimated); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — J591 monoclonal antibody

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- huJ591 followed by 89Zr-J591 (Experimental): Subjects will receive two infusions of unlabeled huJ591 on days 1 and 15 (+/- 1 day). 89Zr-J591 will be administered on day 22 (+/- 1 day) and 5-8 days later. PET/CT will be performed followed by repeat imaging of the prostate. Radical prostatectomy with or without lymph node dissection is performed 2 to 4 weeks after the second dose of J591.
  Interventions: Drug: huJ591; Drug: 89Zr-J591

INTERVENTIONS:
Drug: huJ591 — Antibody is derived from a hybridoma originally produced in the Weill Medical College Laboratory of Urological Oncology. Treatment with 100 mg of HuJ591 will be administered as an intravenous infusion at a concentration of 5 mg/mL and rate of <5 mg/minute.
  Other Names: J591
Drug: 89Zr-J591 — Drug product is manufactured by the radiochemistry staff of Citigroup Biomedical Imaging Center (CBIC) research core facility. Radiolabeling of DFO-huJ591 with 89Zr is achieved by the addition of 89Zr-oxalate to the DFO-huJ591 in ammonium acetate buffer.
  Other Names: radiolabeled J591

SUMMARY:
10 patients will be enrolled in the initial cohort and will receive two infusions of unlabeled huJ591 on days 1 and 14. 89Zr-J591 will be administered on day 21 (+ 1 day) and a positron emission tomography-computed tomography (PET/CT) will be performed week later on day 28 + 1 (visit 4). Approximately 2 to 3 weeks after the 2nd dose of J591, the patient will undergo radical prostatectomy with or without lymph node dissection (day 31 + 4 days). The final visit for the study will include a postoperative visit two weeks following surgery.

DETAILED DESCRIPTION:
This is an open-label, single center pilot study to evaluate the efficacy of huJ591 to trigger antibody-dependent cellular cytotoxicity (ADCC) response manifested by a peri-tumoral inflammatory response with or without apoptosis of prostate cancer cells in patients diagnosed with either high or intermediate-risk prostate cancer. To participate the patients will be required to meet all eligibility criteria. Patients may not participate in other clinical trials while undergoing therapeutic treatment.

The initial screening period (up to 28 days prior to start of treatment under this clinical trial) consists of visit to confirm eligibility, discuss the risks / benefits of participating in the trial and radical prostatectomy (with or without lymph node dissection), and obtain patient prostate biopsy samples for anti-prostate specific membrane antigen (PSMA) expression review. An enrolled subject's participation in the study entails approximately 6 to 7 weeks of therapy along with the additional 2 weeks time involved in recovery from a radical prostatectomy. Adverse events will be collected throughout the entirety of the study. The total duration of the patient being in the study can be around 9 to 11 weeks. Medical information/Survival information will be collected from the routine followup visits (standard of care) for up to 3 years after the surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male > 18 years of age
2. Histologically confirmed diagnosis of prostate cancer
3. Intermediate or high risk prostate cancer defined by:

   * High risk (any one of the following):

     1. Gleason grade > 8
     2. Gleason grade 4+3 with more than 3 cores involved with > 20% of volume involved
     3. Any Gleason with PSA above 20 ng/mL
     4. Gleasone > 4+3 and tumor stage clinical T3 or above
   * Intermediate risk prostate cancer defined as:

     1. Gleason grade = 7
     2. Any Gleason with PSA between 10 and 20 ng/mL
4. Eastern Cooperative Oncology Group (ECOG) Performance status of 0-1
5. Ability to understand and willingness to sign a written informed consent document
6. Prostate biopsy with + PSMA expression in tumor cells by immunohistochemistry

Exclusion Criteria:

1. Serum creatinine > 3x upper limit of normal (ULN)
2. Bilirubin (total) > 1.5 x ULN; subjects with Gilbert's syndrome will be allowed if direct bilirubin is within institutional normal limits
3. Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT or SGOT) > 2.5x ULN
4. Other severe acute or chronic medical condition or laboratory abnormality that may increase the risk associated with study participation
5. On any other new anticancer therapy between screening and prostatectomy
6. Frank metastasis identified during clinical staging
7. Patient ineligible for radical prostatectomy for any other reason

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-02-04 (Actual); Primary Completion 2017-02-10 (Actual); Study Completion 2020-02-02 (Actual)

PRIMARY OUTCOMES:
Induction of inflammatory and/or apoptotic response of prostate cancer cells by reviewing H&E stained slides from pre treatment biopsy and comparing to the post-treatment radical prostatectomy pathology using the Peri-tumoral inflammation 4-point scoring | Change from baseline in Peri-tumoral inflammation 4-point scoring at Day 31 post prostatectomy

SECONDARY OUTCOMES:
Time to biochemical (PSA) and/or radiographic recurrence will be followed by drawing PSA samples and performing radiographic scans. | From date of first treatment until the date of first documented progression or date of death, whichever came first, assessed up to 36 months
  PSA values will be monitored at screening, then at months 3, 6, 9, 12, 18, 24, and 36 after Day 1 of treatment. Radiographic scans will be performed at screening and at months 6, 12, 18, 24, 30, and 36.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Adverse events will be monitored on Days 1, 14, 21, 28, 31, and 45

CONTACTS AND LOCATIONS:
Overall Officials: Scott Tagawa, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No